CLINICAL TRIAL: NCT04297930
Title: Treatment Outcomes of a Novel Glaucoma Tube Shunt Implant for Intraocular Pressure Control in Eyes With Refractory Glaucoma
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/00136
Record Dates: First submitted 2020-02-24; First posted 2020-03-06 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Surgery; Intraocular Pressure
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paul Glaucoma Implant Surgery: Patients who had surgery with the Paul Glaucoma Implant
  Interventions: Device: Paul Glaucoma Implant Surgery

INTERVENTIONS:
Device: Paul Glaucoma Implant Surgery — This group of patients had glaucoma surgery with the Paul Glaucoma Implant

SUMMARY:
The aim of this study is to determine the effectiveness of lowering intraocular pressure and safety profile of the Paul Glaucoma Implant (Advanced Ophthalmic Innovations, Singapore). This is a non-comparative and single-arm observational study and all the participants were recruited between 1 Dec 2017 and 1 Dec 2018. Patients between age 21 - 80 years with glaucoma and an IOP deemed poorly controlled by the study team despite on maximal tolerated medical therapy were included in this study. The participants were recruited from 6 tertiary ophthalmology centers including National University Hospital, Singapore, Moorfields Eye Hospital, United Kingdom, St Thomas' Hospital, United Kingdom, Chulalongkorn University and Hospital, Thailand, International Specialist Eye Centre, Malaysia and Chinese University of Hong Kong, Hong Kong. All the eyes were followed-up for a period of 12 months after surgery. The examination and investigations included best corrected Snellen visual acuity, slit lamp examination, goldman applanation tonometry (GAT), dilated fundus examination and optic nerve head imaging. The participants are reviewed before surgery, 1 day, 1 week, 1 month, three months, 6 months and 12 months after surgery. All the data were captured in a standardized data-collection form for analysis. The primary outcome measure was failure, if was prospectively defined as IOP more than 21mmHg or less than a 20% reduction compared to pre-operative baseline on 2 consecutive visits after 3 months, IOP less than 6 mmHg on 2 consecutive visits after 3 months, reoperation for IOP-related indication, loss of light perception vision, or removal of the implant for any reason. Intraocular pressure outcomes, number of IOP-lowering medications and the rate of surgical complications were secondary outcome measures in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 80 years with glaucoma
* Poorly controlled intraocular pressure

Exclusion Criteria:

* Unable to give informed consent
* Age below 21 or above 80 years
* Without any suitable quadrants for tube shunt implant

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between age 21 - 80 years with glaucoma and an IOP deemed poorly controlled by the study team despite on maximal tolerated medical therapy were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 12 months
  The primary outcome measure was surgical failure, if was prospectively defined as IOP more than 21mmHg or less than a 20% reduction compared to pre-operative baseline on 2 consecutive visits after 3 months, IOP less than 6 mmHg on 2 consecutive visits after 3 months, reoperation for IOP-related indication, loss of light perception vision, or removal of the implant for any reason

SECONDARY OUTCOMES:
Number of intraocular-pressure-lowering medications | 12 months
  Complete success was defined as IOP less than or equal to 21 mmHg and more than 5 mmHg, IOP reduced by more than or equal to 20% from baseline and medications were not used at either the 6 or 12 month visits
  Qualified success is similarly defined but with the use of IOP-lowering medications. In addition, we also provided success rates based on alternative upper limit of IOP at 18 and 15 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Victor Koh, MBBS, MMed, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No